CLINICAL TRIAL: NCT06485219
Title: An Open-Label, Multicenter Phase IIa Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Purinostat Mesylate for Injection for the Treatment of Patients With Relapsed or Refractory Peripheral T-Cell Lymphoma and Cutaneous T-Cell Lymphoma
Brief Title: A Phase IIa Clinical Study of Purinostat Mesylate for Injection in Patients With Peripheral T-Cell Lymphoma and Cutaneous T-Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chengdu Zenitar Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZLPM-004-1.0
Record Dates: First submitted 2024-05-22; First posted 2024-07-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Relapsed or Refractory Peripheral T-cell Lymphoma (PTCL); Cutaneous T-cell Lymphoma (CTCL)
MeSH Terms: conditions — Recurrence; Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 11.2mg/m2 Purinostat Mesylate group (Experimental)
  Interventions: Drug: 11.2 mg/m2 Purinostat Mesylate
- 15.0mg/m2 Purinostat Mesylate group (Experimental)
  Interventions: Drug: 15 mg/m2 Purinostat Mesylate

INTERVENTIONS:
Drug: 11.2 mg/m2 Purinostat Mesylate — Purinostat Mesylate for Injection: Intravenous infusion, The subjects were given intravenous drip injections once on D1, D4, D8 and D11 of each dosing cycle, with a dosing cycle lasting for 21 days. The overall duration of the longest administration period shall not exceed 96 weeks.
  Arms: 11.2mg/m2 Purinostat Mesylate group
Drug: 15 mg/m2 Purinostat Mesylate — Purinostat Mesylate for Injection: Intravenous infusion, The subjects were given intravenous drip injections once on D1, D4, D8 and D11 of each dosing cycle, with a dosing cycle lasting for 21 days. The overall duration of the longest administration period shall not exceed 96 weeks.
  Arms: 15.0mg/m2 Purinostat Mesylate group

SUMMARY:
Primary Objective To evaluate the preliminary efficacy of Purinostat Mesylate for Injection in patients with relapsed or refractory Peripheral T-Cell Lymphoma (PTCL) and Cutaneous T-Cell Lymphoma (CTCL).

Secondary Objectives

1. To evaluate the safety and tolerability of Purinostat Mesylate for Injection in patients with relapsed or refractory PTCL and CTCL.
2. To evaluate the population pharmacokinetic characteristics of Purinostat Mesylate for Injection in patients with relapsed or refractory PTCL and CTCL.

Exploratory Objective To investigate the relationship between tumor biomarkers and the therapeutic efficacy/safety profile of Purinostat Mesylate for Injection.

ELIGIBILITY:
Inclusion Criteria:

1. The patient fully understands this study, voluntarily participates, and signs the informed consent form (ICF). They are able to communicate well with the investigator and can adhere to the study's visit schedule, treatment plan, laboratory tests, and other study procedures.
2. Aged ≥18 years, male or female;
3. Histologically confirmed diagnosis based on the 2022 revised World Health Organization (WHO) classification criteria, including but not limited to the following subtypes:

   1. Peripheral T-cell lymphoma, not otherwise specified (PTCL-NOS),
   2. NK/T-cell lymphoma (nasal type),
   3. Angioimmunoblastic T-cell lymphoma (AITL),
   4. Anaplastic large cell lymphoma (ALCL),
   5. Enteropathy-associated T-cell lymphoma (EATL),
   6. Hepatosplenic T-cell lymphoma (HSTL),
   7. Cutaneous T-cell lymphoma at TNMB stage IB-IVA,
   8. Other subtypes of PTCL that the investigator considers eligible and are approved by the sponsor (excluding highly aggressive subtypes).
4. Prior treatment: Relapsed/refractory PTCL refers to patients who have failed or are intolerant to at least one line of systemic standard treatment (≤5 lines). For NK/T-cell lymphoma, prior treatment must include asparaginase/pegaspargase/L-asparaginase. For other subtypes, prior treatment must include anthracyclines (unless anthracyclines are contraindicated).Relapsed/refractory CTCL refers to patients who have relapsed, progressed, or were unresponsive after adequate treatment with at least one systemic therapy (e.g., interferon, retinoids).The detailed definitions of relapsed/refractory PTCL are as follows: Relapse: Refers to disease progression after achieving remission (including complete remission and partial remission) with prior first-line treatment. This includes: a) Completion of treatment according to clinically recommended standards or conventional regimens (for early-stage patients, combined chemoradiotherapy with at least 2 cycles of recommended chemotherapy; for advanced-stage patients, systemic treatment with at least 4 cycles for those who received hematopoietic stem cell transplantation consolidation, or at least 6 cycles for those who did not).

   b) Relapse within 1-3 years after remission, and not suitable for or unwilling to undergo autologous hematopoietic stem cell transplantation salvage therapy.

   Refractory: Refers to patients who did not achieve remission with prior first-line treatment or experienced disease progression during treatment or within 1 year after completing treatment. This includes:a) Failure to achieve stable disease (SD) after ≥2 cycles of treatment according to clinically recommended standards or conventional regimens, or failure to achieve partial remission (PR) after ≥3-4 cycles.b) If the best response or reason for ending treatment was progressive disease (PD), the number of treatment cycles is not required.

   c) Disease progression after receiving ≥2 lines of clinically recommended standard or conventional treatment. d) Relapse after autologous hematopoietic stem cell transplantation.
5. Expected survival > 3 months.
6. ECOG score 0-2.
7. Patients with PTCL have at least one measurable lesion according to the 2014 Lugano criteria (lesions that have received radiotherapy can be used as target lesions if there is clear evidence of disease progression after radiotherapy), with a measurable lesion defined as: an intranodal lesion with a maximum diameter of >1.5 cm on CT cross-sectional images; or an extranodal lesion with a maximum diameter of >1.0 cm; patients with CTCL must have an mSWAT score ≥10% with or without systemic lymph node invasion;
8. Organ function levels must meet the following requirements: routine blood tests (no growth factors or blood transfusions within 14 days prior to screening): absolute neutrophil count (ANC) ≥1.0×10^9/L; hemoglobin (HGB) ≥80 g/L; platelet count (PLT) ≥75×10^9/L (patients with bone marrow infiltration of lymphoma ≥50×10^9/L can be enrolled); liver and kidney function: serum ≥10%, serum ≥10%, serum ≥50×10^9/L (patients with bone marrow infiltration of lymphoma ≥50×10^9/L). ); liver and kidney function: serum total bilirubin ≤1.5 × upper limit of normal (ULN) (TBiL ≤3.0 × ULN in patients with Gilbert's syndrome may be enrolled); aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤2.5 × ULN, or in the judgment of the investigator, when there is hepatic infiltration resulting in hepatic function impairment. ALT, AST, and ALP ≤ 5 × ULN may be enrolled; serum creatinine ≤ 1.5 × ULN or estimated creatinine clearance ≥ 50 mL/min (according to the Cockcroft and Gault formula); coagulation: activated partial thromboplastin time (APTT), International Normalized Ratio (INR), and prothrombin time (PT) ≤ 1.5 × ULN, and Fibrinogen (FIB) ≥ 1.0 g/L;
9. Females and males of childbearing potential should agree that effective contraception (hormonal or barrier methods or abstinence) is required during the study and for 6 months after study completion; female patients of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to administration of the drug and must be non-lactating.

Exclusion Criteria:

1. Patients with leukemic PTCL (e.g., adult T-cell leukemia/lymphoma, etc.), or lymphomatous leukemia stage (percentage of lymphoma cells ≥20% on bone marrow examination), or central nervous system (CNS) involvement, or concomitant hemophagocytic syndrome;
2. Have a history of allergy to similar drugs and excipients of the test drug;
3. Have received any other antitumor therapy [including chemotherapy with cytotoxic agents, molecularly targeted therapy, immunotherapy, or other biological therapies within 4 weeks prior to the first use of the test drug, mitomycin or nitrosamines within 6 weeks, small molecule targeted agents at least 2 weeks or at least 5 half-life intervals from the last dose, whichever is longer, and traditional Chinese medicines with antitumor indications at least 2 weeks from the last dose], and have received the test drug within 4 weeks prior to the first use of the test drug, or have a history of hypersensitivity to similar drugs and excipient components of the test drug; or have a history of allergy to the test drug. Chinese herbal medicines with antitumor indications should be administered at least 2 weeks after the last dose], and local radiotherapy within 4 weeks prior to the first administration of the test drug;
4. The presence of persistent Grade 2 or above (CTCAE V5.0 standard) toxicity reaction after the previous treatment (chemotherapy or biotherapy or targeted therapy, etc.), which has not yet recovered to Grade ≤1 level at the time of enrollment (with the exception of alopecia areata);
5. Vaccination with live attenuated vaccine within 28 days prior to the first dose of study drug or within 60 days of the end of treatment with study drug;
6. Have received a blood transfusion, recombinant human thrombopoietin, erythropoietin, or granulocyte colony-stimulating factor within 2 weeks prior to the first dose of the investigational drug;
7. A history of solid organ or allogeneic hematopoietic stem cell transplantation; autologous hematopoietic stem cell transplantation within 3 months prior to the first dose of the investigational drug;
8. Patients who have received any of the following treatments within 7 days prior to the first dose of the investigational drug: drugs known to be potent inhibitors/inducers of CYP 3A4, drugs known to significantly prolong the QT period;
9. Uncontrolled electrolyte disturbances that may interfere with the action of QTc prolonging medications (e.g., hypocalcemia <1.0 mol/L, hypokalemia <lower limit of normal, hypomagnesemia <0.5 mmol/L), but retesting after interventional therapy is permitted;
10. Major surgery (other than tumor biopsy) within 4 weeks prior to the first trial drug administration, or the patient has not recovered and the side effects of the surgery have not stabilized;
11. Presence of uncontrolled Grade 2 or higher (CTCAE V5.0 criteria) active clinical infection requiring systemic anti-infective treatment (except if the patient's infection has been controlled and anti-infective treatment still needs to be maintained);
12. Treatment with prednisone >10 mg/day [CTCL >20 mg/d (equivalent prednisone dose)] within 7 days prior to the first dose of the test drug, except for the following: treatment with topical, ophthalmic, intra-articular, intranasal, and inhaled corticosteroids, short-term prophylactic corticosteroid use for Treatment, e.g., with contrast media;
13. Impaired cardiac function or significant cardiac disease, including but not limited to:

1) Myocardial infarction, congestive heart failure, viral myocarditis within 6 months prior to screening; symptomatic requiring therapeutic intervention for heart disease, such as unstable angina, arrhythmia, etc; 2) Cardiac function class III to IV (New York Heart Association cardiac function classification NYHA); 3)Left ventricular ejection fraction (LVEF) of less than 50% by cardiac radionuclide scanning (MUGA) or echocardiography (ECHO) or less than the lower limit of the laboratory test value at the research center; 4) History of persistent cardiomyopathy, primary cardiomyopathy (e.g., dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, and undetermined cardiomyopathy); 5) Screening-phase symptomatic coronary heart disease requiring pharmacologic treatment; 6) A history of clinically significant QTcF interval prolongation or a mean corrected QT interval (QTcF) >450 msec (men) or >470 msec (women) on 3 electrocardiograms (ECGs) at rest during the screening period (retesting is required only if the first ECG suggests a QTcF of >450 msec (men) or >470 msec (women)) and is taken at a later date. 3 average corrected values); history of or confirmed family history of long QT syndrome; history of clinically significant ventricular arrhythmia or current use of antiarrhythmic drugs or implanted defibrillation device for the treatment of ventricular arrhythmias; 14. Cerebrovascular accident (including transient ischemic attack or symptomatic pulmonary embolism) within 6 months prior to screening; 15. patients with uncontrolled hypertension (defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥95 mmHg after standardized antihypertensive treatment) or diabetes mellitus with poor glycemic control (random blood glucose ≥13.9 mmol/L after hypoglycemic treatment, or HbA1c ≥8.5%) 16. A history of hepatic fibrosis or cirrhosis, or clinical signs and symptoms suggestive of hepatic fibrosis or cirrhosis. Severe lung disease (CTCAE V5.0 Class III-IV); 17. Presence of third interstitial fluid (e.g., massive pleural fluid and ascites) that cannot be controlled by drainage or other means.

18. Combination of any other malignancy (adequately treated and effectively controlled non-melanotic cutaneous basal cell or cutaneous squamous epithelial cell carcinoma or cervical carcinoma in situ, carcinoma in situ of the breast/cervix, superficial bladder cancer, limited prostate cancer, other appropriately treated stage 1 or stage 2 cancer in complete remission, or any other cancer in complete remission).

Hepatitis B virus (HBV) (except Stage 1 or Stage 2 cancers in complete remission, or any other cancer that has been in complete remission for more than 5 years); known or existing primary or metastatic central nervous system lymphomas and subjects with symptomatic brain metastases; 19. Active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV), except for the following patients: a) HBV infection: Hepatitis B surface antigen (HbsAg) or Hepatitis B core antibody (HbcAb) positivity, and then peripheral blood Hepatitis B DNA titer test, HBV DNA ≤ 1 x 103 copies/ml (or the lower limit of the assay value) can be enrolled; after enrollment, a holders' license is required. Patients with HBV DNA ≤1×103 copies/ml (or the limit of detection) can be enrolled; after enrollment, they need to continue antiviral treatment and have hepatitis B DNA titer test every cycle; b) Patients with positive HCV serology but negative HCV RNA test can be enrolled. Patients who are seropositive for HCV but negative for HCV RNA may be enrolled.

Antibody (HIV-Ab) or anti-syphilis spirochete antibody (TP-Ab) positive ; 20. History of psychiatric illness, family history of psychiatric illness, or mood disorders as determined by the investigator or psychologist [including medically documented history of depressive episodes, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, suicidal attempts or suicidal ideation, or homicidal ideation (immediate risk of harm to others)].

history of suicide attempts or suicidal ideation, or homicidal ideation (immediate risk of harm to others), anxiety level 3 or higher, etc.]; 21. Participation in another clinical study and treatment with the trial drug within 4 weeks prior to the first dose of trial drug; 22. Any condition that, in the judgment of the investigator, is unstable or may jeopardize the safety of the subject and his/her compliance with the study; 23. Any other factors that, in the opinion of the investigator, make participation in the trial inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate (ORR) | Evaluated every two cycles (Each cycle is 21 days)
  Defined as the proportion of subjects with an overall efficacy response of complete remission (CR) or partial remission (PR) after at least one post-baseline evaluation during the trial period

SECONDARY OUTCOMES:
Complete Remission Rate (CRR) | Evaluated every two cycles (Each cycle is 21 days)
  Defined as the proportion of subjects with an overall efficacy response of CR after at least one post-baseline evaluation during the trial;
Disease Control Rate (DCR) | Evaluated every two cycles (Each cycle is 21 days)
  Defined as the proportion of subjects with an overall efficacy response of CR, PR, and stable disease (SD) after at least one post-baseline evaluation during the trial;
Duration of remission (DOR) | Evaluated every two cycles (Each cycle is 21 days)
  Duration of first remission (PR or CR) to disease progression or death;
Time to Tumor Remission (TTR) | Evaluated every two cycles (Each cycle is 21 days)
  Time from first dose to the onset of remission
Progression-Free Survival (PFS) | Week 96
  Defined as the time from the first administration of the drug to disease progression or death (whichever occurs first).
Overall Survival (OS) | Week 96
  Defined as the time from the first administration of the drug to death (due to any cause).

CONTACTS AND LOCATIONS:
Overall Officials: Ting Niu, Doctor, Principal Investigator — West China Hospital; Weili Zhao, Doctor, Principal Investigator — Ruijin Hospital
Locations (2):
- China (2):
  - Ruijin Hospital, Shanghai Jiaotong University School Of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No